CLINICAL TRIAL: NCT04753801
Title: What Are the Ingredients for the Best Form of the Best Possible Self (BPS) Intervention? Combining the BPS Intervention With Mindfulness
Brief Title: What Are the Ingredients for the Best Form of the Best Possible Self (BPS) Intervention?
Acronym: BestBPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BestBPS
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Best Possible Self (writing only) (Experimental): Participants are asked to think and write about their best possible future self (15 min).
  Interventions: Behavioral: Thinking, writing and imagination
- Best Possible Self (writing+imagining) (Experimental): Participants are asked to think and write about their best possible future self (15 min) and, then to imagine their positive future (5 min).
  Interventions: Behavioral: Thinking, writing and imagination
- Best Possible Self (writing+mindfulness) (Experimental): Participants are asked to think and write about their best possible future self (15 min) and subsequently engage in a brief mindfulness sequence (5 min).
  Interventions: Behavioral: Thinking, writing and imagination
- Best Possible Self (writing+recall) (Experimental): Participants are asked to think and write about their best possible future self (15 min) and subsequently engage in a brief recall imagination task about the past two days (5 min).
  Interventions: Behavioral: Thinking, writing and imagination
- Writing about the past (Active Comparator): Participants are asked to think and write about activities of the past two days (15 min).
  Interventions: Behavioral: Thinking, writing and imagination

INTERVENTIONS:
Behavioral: Thinking, writing and imagination — All participants are asked to take some time to think and write about the respective intervention group's content. In some groups (after the writing exercise (approx. 15min)), participants are also asked to imagine that content or engage in a mindfulness activity or recall task for about 5 minutes.

SUMMARY:
This study aims to determine the relevant 'ingredients' to make the best possible self (BPS) intervention most efficacious and test whether the BPS's efficacy can be enhanced by including mindfulness aspects.

DETAILED DESCRIPTION:
The best possible self (BPS) intervention is a brief positive psychology intervention to increase a person's positive affect and optimism. The BPS has been used in different forms (writing vs. imagining/visualizing vs. writing + imagining/visualizing the best possible self). However, it remains unclear which 'ingredients' are necessary to let the BPS unfold its effects. This online study aims to determine the relevant 'ingredients' to make the best possible self (BPS) intervention most efficacious. Since mindfulness interventions have recently indicated promising effects on positive and negative affect, another goal of this study is to test whether the BPS's efficacy can be enhanced by including aspects of mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* fluent in the German language
* access to a computer/tablet/smartphone with audio output/headphones

Exclusion Criteria:

* not willing to take part in an online-intervention (duration: 60 minutes)
* no access to a computer/tablet/smartphone with audio output/headphones

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in emotions (PANAS) | Change from pre (baseline) to post scores (approx. 30 minutes later)
  Change scores are calculated for positive and negative sum scores (post- minus pre-scores; pre-scores will be used as a covariate).

SECONDARY OUTCOMES:
Change in state optimism ratings | Change from pre (baseline) to post scores (approx. 30 minutes later)
  State Optimism measure (SOM), 7 items (each item 1(strongly disagree)-5(strongly agree)). Change scores are calculated for positive and negative sum scores (post- minus pre-scores; pre-scores will be used as a covariate).
Change in emotional responses to imagery of neutral, pleasant and aversive narrative scripts | Change from pre (baseline) to post scores (approx. 30 minutes later)]
  Nine narrative imagery scripts are used. Scenes included three neutral, standard social threat and positive/reward events. All scripts were developed according to the recommendations of Lang (1979). Participants are asked to rate the vividness of imagery (1= not vivid at all, 9= very vivid), the wish to avoid imagery (1 = no wish to avoid , 9 = strong wish to avoid imagery), their experienced anxiety (1= no anxiety, 9=very strong anxiety), displeasure (1 = pleasant, 9 = unpleasant), and emotional arousal (1 = relaxed, 9 = aroused) during imagery on a 9-point rating scale. Emotional responses are averaged per category.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof., Principal Investigator — Philipps University Marburg
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data will be shared with researchers providing a relevant and methodologically sound proposal

REFERENCES:
- [Background] Millstein RA, Chung WJ, Hoeppner BB, Boehm JK, Legler SR, Mastromauro CA, Huffman JC. Development of the State Optimism Measure. Gen Hosp Psychiatry. 2019 May-Jun;58:83-93. doi: 10.1016/j.genhosppsych.2019.04.002. Epub 2019 Apr 4. PMID 31026732